CLINICAL TRIAL: NCT06913608
Title: A Phase lb Open-Label Study Evaluating the Safety and Efficacy of the Combination of CLBR00l, an Engineered Autologous T Cell Product, and SWI019, a CD19-directed Antibody-based Biologic With or Without Lymphodepletion in Subjects With Autoimmune Disorders Including Systemic Lupus Erythematosus, Systemic Sclerosis, or Idiopathic Inflammatory Myositis
Brief Title: A Study to Assess CLBR001+SWI019 in Subjects With Autoimmune Diseases
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Calibr, a division of Scripps Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBR-sCAR19-3003
Record Dates: First submitted 2025-03-28; First posted 2025-04-06 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erythematosus (SLE); Systemic Sclerosis (SSc); Idiopathic Inflammatory Myopathy (IIM)
Keywords: CAR-T; systemic lupus erythematosus; systemic sclerosis; idiopathic inflammatory myopathy; SLE; IIM; SSc; cell therapy
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Scleroderma, Systemic; Myositis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CLBR001 + SWI019 following Lymphodepletion (Experimental): Subjects who are randomized into the lymphodepletion arm will undergo 3 days of lymphodepletion conditioning therapy consisting of fludarabine and cyclophosphamide prior to treatment with CLBR001+SWI019.
  Interventions: Combination Product: CLBR001 + SWI019
- CLBR001 + SWI019 without Lymphodepletion (Experimental): Subjects who are randomized into the NO lymphodepletion arm will receive treatment with CLBR001+SWI019 without lymphodepletion administered prior.
  Interventions: Combination Product: CLBR001 + SWI019

INTERVENTIONS:
Combination Product: CLBR001 + SWI019 — Investigational switchable CAR-T cell therapy for autoimmune disorders

SUMMARY:
The goal of this clinical trial is to evaluate CLBR001 and SWI019 as a treatment for patients with autoimmune disorders, including systemic lupus erythematosus, systemic sclerosis, and idiopathic inflammatory myositis. Patients will be randomized 1:1 lymphodepletion vs no lymphodepletion arm. Patients will be administered a single infusion of CLBR001 cells followed by cycles of SWI019 with regular assessments of safety and disease response to treatment.

The goals are to establish the safety and efficacy of the combination therapy and determine if lymphodepletion is required for efficacy.

DETAILED DESCRIPTION:
CLBR001 + SWI019 is novel switchable CAR-T cell combination therapy comprised of an autologous CAR (chimeric antigen receptor)-T product (CLBR001, the switchable CAR-T cell [sCAR-T]) and SWI019 (the "switch" biologic molecule). SWI019 acts as an adapter molecule that controls the activity of the CLBR001 CAR-T cell product.

ELIGIBILITY:
Inclusion Criteria:

* Women or men age ≥18 of age at time of consent.
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of this study.
* Adequate hematological, liver, pulmonary, and cardiac function
* Willing to participate to participate in long term follow up study.
* Confirmed diagnosis of moderate to severe systemic lupus erythematosus with lupus nephritis, systemic lupus erythematosus with extrarenal lupus, systemic sclerosis, and idiopathic inflammatory myositis.
* Failed at least two immunosuppressive treatments

Exclusion Criteria:

* Inability to tolerate washout of prior therapy.
* Not willing/understanding the requirements of the clinical study
* Dependent on hemodialysis for a period of greater or equal to 3 months.
* Known hypersensitivity to prednisone or to both tocilizumab siltuximab.
* Have received plasmapheresis within 14 days prior to informed consent.
* Active bacterial, viral and/or fungal infection.
* Prior autologous/allogeneic stem cell transplant or solid organ transplant.
* Prior lentiviral or retroviral based therapy including CAR-T cell therapy.
* History or concurrent malignancy with active treatment in the past 5 years
* HIV-1 and HIV-2 antibody positive subjects.
* History of central nervous system diseases (such as seizure, psychosis, organic brain syndrome or cerebrovascular accident).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with adverse events | To 1 year post CLBR001 administration
  To assess the safety and tolerability in subjects by evaluating the frequency, relatedness, severity and duration of adverse events (assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0, with exception of Cytokine Release Syndrome (CRS) or Immune effector Cell-Associated Neurotoxicity Syndrome (ICANS) which will be graded by American Society for Transplantation and Cellular Therapy (ASTCT) consensus grading criteria).

SECONDARY OUTCOMES:
Evaluate the efficacy of CLBR001 + SWI019 in autoimmune disease | 1 year post CLBR001 administration
  Efficacy will be measured by the number of subjects with a clinical response.
Quantification of white blood cells (WBCs) | 1 year post CLBR001 administration
  Quantify WBCs, i.e. monocytes, neutrophils, other granulocytes, and lymphocytes, in peripheral blood to evaluate changes in circulating WBCs between subjects assigned to lymphodepletion vs no lymphodepletion arms to determine role of lymphodepletion in CAR-T cell engraftment.
Evaluate the pharmacokinetics (PK) of CLBR001 and SWI019: Maximum Concentration (Cmax) | 1 year post CLBR001 administration
  Quantitation and persistence of CLBR001 cells in peripheral blood and PK parameters of SWI019
Assess immunogenicity of CLBR001 and SWI019 | 1 year post CLBR001 administration
  Immunogenic response to CLBR001 and SWI019 will be measured by presence of antidrug antibodies (ADA).
Number of subjects with Clinical Response | 1 year post CLBR001 administration
  Evaluate anti-disease activity of CLBR001 and SWI019 by number of subjects with Clinical Response to treatment.
Evaluate the pharmacokinetics (PK) of CLBR001 and SWI019: Time to Peak Drug Concentration (Tmax) | 1 year post CLBR001 administration
  Quantitation and persistence of CLBR001 cells in peripheral blood and PK parameters of SWI019
Evaluate the pharmacokinetics (PK) of CLBR001 and SWI019: Area Under the Curve (AUC) | 1 year post CLBR001 administration
  Quantitation and persistence of CLBR001 cells in peripheral blood and PK parameters of SWI019
Evaluate the pharmacokinetics (PK) of CLBR001 and SWI019: Half-life (t1/2) | 1 year post CLBR001 administration
  Quantitation and persistence of CLBR001 cells in peripheral blood and PK parameters of SWI019

CONTACTS AND LOCATIONS:
Overall Officials: Calibr CMO, Study Director — Calibr-Skaggs, Institute of Innovative Medicines

IPD SHARING:
Plan to Share IPD: No